CLINICAL TRIAL: NCT00771849
Title: Antibody Responses for Serogroup C After One Dose of an Experimental Tetravalent (A, C, Y, and W-135) Meningococcal Diphtheria Toxoid Conjugate Vaccine Versus a Non-meningococcal Control Vaccine in Children Who Have Previously Received a Monovalent Meningococcal C Conjugate Vaccine
Brief Title: Study of Antibody Responses After a Dose of Tetravalent Meningococcal Diphtheria Conjugate Vaccine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTA15
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2009-04-24 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Meningitis; Meningococcemia
Keywords: Meningitis; Meningococcemia; Neisseria meningitidis
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines; Vaccines; Hiberix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Menactra® Vaccine Group (Experimental): Participants receiving the tetravalent (A, C, Y, and W 135) meningococcal diphtheria toxoid conjugate vaccine
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Hiberix® Vaccine Group (Active Comparator): Participants receiving Haemophilus Influenzae Type b (Hib) vaccine
  Interventions: Biological: Haemophilus Influenzae Type b (Hib) vaccine

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Vaccine Group
Biological: Haemophilus Influenzae Type b (Hib) vaccine — 0.5 mL, Intramuscular
  Other Names: Hiberix®
  Arms: Hiberix® Vaccine Group

SUMMARY:
The study investigated safety profile and the antibody responses to an experimental tetravalent meningococcal diphtheria conjugate vaccine (Menactra®) in children who have received a monovalent meningococcal C conjugate vaccine at least one year previously.

Primary objective:

To describe and compare the Serum Bactericidal Assay (SBA) antibody response for serogroup C in participants receiving Menactra® to the serogroup C antibody response in a control group of participants receiving a licensed Haemophilus Influenzae Type b (Hib) conjugate vaccine 28 days following vaccination.

ELIGIBILITY:
Inclusion Criteria :

* Participant is healthy, as determined by medical history and physical examination.
* Participant is 2 years to < 5 years of age at the time of vaccination.
* At least one year from primary vaccination with a monovalent meningococcal C conjugate vaccine has elapsed.
* Parent/Guardian has signed an Ethics Committee-approved informed consent form. A culturally appropriate translation will be used for non-English speaking participants where required.

Exclusion Criteria :

* Serious chronic disease (i.e. cardiac, renal, neurologic, metabolic, rheumatologic, etc.)
* Known or suspected impairment of immunologic function
* Acute medical illness with or without fever within the last 72 hours or an axillary temperature ≥ 37.5ºC at the time of inclusion
* History of documented invasive meningococcal disease
* Administration of immune globulin, other blood products within the last three months, injected or oral corticosteroids or other immunomodulatory therapy within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrolment
* Antibiotic therapy within the 72 hours prior to vaccination or 72 hours prior to drawing any blood sample
* Received any vaccine in the 28-day period prior to enrolment, or scheduled to receive any vaccine during enrolment in the trial
* Received a meningococcal C conjugate vaccine within one year prior to enrolment
* Suspected or known hypersensitivity to any of the vaccine components
* Unavailable for the entire study period or unable to attend the scheduled visits or to comply with the study procedures
* Enrolled in another clinical trial
* Any condition, which, in the opinion of the investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2003-08; Primary Completion 2004-03 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (1):
- London, United Kingdom

REFERENCES:
- [Result] El Bashir H, Heath PT, Papa T, Ruggeberg JU, Johnson N, Sinha R, Balfour G, Booy R. Antibody responses to meningococcal (groups A, C, Y and W135) polysaccharide diphtheria toxoid conjugate vaccine in children who previously received meningococcal C conjugate vaccine. Vaccine. 2006 Mar 24;24(14):2544-9. doi: 10.1016/j.vaccine.2005.12.018. Epub 2005 Dec 27. PMID 16417952
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from August 2003 through March 2004 at 2 clinics in the United Kingdom.
Pre-assignment Details: A total of 103 subjects that met the inclusion but none of the exclusion criteria were enrolled, 102 subjects were vaccinated.
Groups:
- Menactra® Vaccine Group: Participants received Menactra® Vaccine
- Hiberix® Vaccine Group: Participants received Hiberix® Vaccine
Period: Overall Study
Arm/Group | Menactra® Vaccine Group | Hiberix® Vaccine Group
Started | 52 | 51 (One subject was not vaccinated)
Completed | 50 | 47
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Not vaccinated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menactra® Vaccine Group | Hiberix® Vaccine Group | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52 | 51 | 103
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 37.0 (8.5) | 37.6 (8.3) | 37.3 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 22 | 50
  Male | 24 | 29 | 53
Region of Enrollment [Number; unit: participants]
  United Kingdom | 52 | 51 | 103

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean of Antibody Titers (GMTs) as Measured by Serum Bactericidal Assay (SBA) at Baseline (Day 0) and Day 28 Post-vaccination.
Time Frame: Day 0 (before) and 28 days post-vaccination
Population: SBA geometric mean titers for each of the 4 meningococcal serogroups was evaluated in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Menactra® Vaccine Group | Hiberix® Vaccine Group
Number analyzed (Participants) | 44 | 36
Titers
  Meningococcal Serogroup A - Day 0 | 136.33 [69.39 to 267.84] | 99.66 [47.66 to 208.40]
  Meningococcal Serogroup A - Day 28 | 11404.16 [7383.63 to 17613.96] | 199.31 [93.14 to 426.52]
  Meningococcal Serogroup C - Day 0 | 76.11 [36.57 to 158.41] | 26.91 [12.49 to 57.97]
  Meningococcal Serogroup C - Day 28 | 12534.67 [8407.56 to 18687.71] | 22.63 [10.50 to 48.76]
  Meningococcal Serogroup Y - Day 0 | 236.61 [133.11 to 420.60] | 266.05 [151.05 to 468.59]
  Meningococcal Serogroup Y - Day 28 | 4031.98 [2399.10 to 6776.24] | 298.63 [155.64 to 572.99]
  Meningococcal Serogroup W-135 - Day 0 | 26.07 [13.30 to 51.13] | 24.44 [11.76 to 50.79]
  Meningococcal Serogroup W-135 - Day 28 | 5978.03 [3852.54 to 9276.19] | 32 [16.33 to 62.71]

2. Secondary Outcome: Participants With a ≥ 4-Fold Rise in Antibody Titers as Measured by Serum Bactericidal Assay (SBA) From Baseline to Day 28 Post-vaccination.
Time Frame: 28 days post-vaccination
Population: SBA titers for each of the 4 meningococcal serogroups was evaluated in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group | Hiberix® Vaccine Group
Number analyzed (Participants) | 44 | 36
Participants
  Meningococcal Serogroup A | 43 | 11
  Meningococcal Serogroup C | 41 | 2
  Meningococcal Serogroup Y | 35 | 1
  Meningococcal Serogroup W-135 | 43 | 8

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 28 days post-vaccination.
Description: One participant in the Menactra® vaccine group and 3 participants in the Hiberix® vaccine group that did not complete the study also did not report any unsolicited adverse event.
Arm/Group | Menactra® Vaccine Group | Hiberix® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/50
Other Adverse Events (participants affected / at risk) | 15/52 | 22/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra® Vaccine Group (N=52) | Hiberix® Vaccine Group (N=50)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Menactra® Vaccine Group (N=52) | Hiberix® Vaccine Group (N=50)
Diarrhoea NOS (Gastrointestinal disorders) | 2/51 | 3/47
Pyrexia (Gastrointestinal disorders) | 1/51 | 3/47
Gastroenteritis NOS (Infections and infestations) | 0/51 | 3/47
Otitis media NOS (Infections and infestations) | 0/51 | 3/47
Upper respiratory tract infection NOS (Infections and infestations) | 10/51 | 14/47
Cough (Respiratory, thoracic and mediastinal disorders) | 3/51 | 3/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.